CLINICAL TRIAL: NCT02051231
Title: Recovery of Oxytocin Responsiveness in Pregnant Human Myometrial Explants After Oxytocin-Induced Desensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-01
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Oxytocin receptors; Oxytocin desensitization
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): A control sample from each patient (no oxytocin applied) will be measured concurrently with samples treated with oxytocin.
- Oxytocin (Experimental): Samples from each patient will be exposed to oxytocin and then allowed to rest for 30, 60 or 90 minutes.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-10mol/L to 10-5mol/L
  Other Names: Pitocin
  Arms: Oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal morbidity and mortality worldwide and is caused most commonly by poor uterine muscle tone after delivery. The first line agent used in the prevention and treatment of PPH is oxytocin, which acts by binding with oxytocin receptors (OTR) found on myometrial cells to cause uterine contraction.

Women who require augmentation of labour with oxytocin because of inadequate labour progression are at increased risk of PPH because they have received intravenous oxytocin which exposes the uterus (and OTR) to doses greater than would normally be found without medical intervention. This exposure results in OTR desensitization and decreased uterine sensitivity to oxytocin which may lead to the use of much higher doses of oxytocin (up to 9x) or other agents for preventing and treating PPH with the potential for causing serious drug-related morbidity or fatality to the mother.

Currently, in women who have failed labour augmentation and need to have a Cesarean delivery, it is not known if it would be beneficial to wait a certain period of time after discontinuing intravenous oxytocin before proceeding with the operation. The goal of the waiting time would be to allow the OTRs to recover and resensitize the uterus to the effects of oxytocin to avoid the need for high doses or additional uterus-contracting agents.

Our hypothesis is that there will be a positive correlation between the magnitude of recovery of the myometrium's response to oxytocin and the time elapsed from the desensitizing oxytocin pretreatment (simulated labour augmentation).

DETAILED DESCRIPTION:
The investigators have previously established an in vitro model of labour augmentation and myometrial desensitization using pregnant human myometrium and an isometric tension recording device. The investigators propose to use this model in order to characterize the time course of recovery of oxytocin-desensitized myometrium to oxytocin sensitivity. These results will help in establishing whether myometrial recovery can occur within a clinically relevant time period, how much sensitivity is recovered, and the duration required.

In the clinical setting of failed labour augmentation and OTR desensitization, it is not known if it is beneficial to wait a certain period of time after discontinuing intravenous oxytocin before proceeding to Cesarean section to allow for resensitization of the myometrium to oxytocin. The results of this study will provide insight into the time course of recovery of the myometrium using an in vitro model of failed labour augmentation. Based on the oxytocin dose-response curves after variable periods of time of "rest", the investigators will be able to determine the degree of recovery of myometrial contractility over time and whether this will occur in a clinically relevant time period for implementation into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who give written consent to participate in this study
* Patients with gestational age 37-41 weeks
* Non-laboring patients, not exposed to exogenous oxytocin
* Patients requiring primary Cesarean section or first repeat Cesarean section

Exclusion Criteria:

* Patients who refuse to give written informed consent
* Patients who require general anesthesia
* Patients who had previous uterine surgery or more than one previous Cesarean section
* Patients with a multiple pregnancy (more than one fetus)
* Patients with any condition predisposing to uterine atony and postpartum hemorrhage, such as abnormal placentation, multiple gestation, preeclampsia, macrosomia, polyhydramnios, uterine fibroids, bleeding diathesis, chorioamnionitis, or a previous history of postpartum bleeding
* Emergency Cesarean section in labor
* Patients with bleeding disorders

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Amplitude of contraction | 2-4 hours

SECONDARY OUTCOMES:
frequency of contraction | 2-4 hours
Integrated area under response curve (AUC) | 2-4 hours
basal tone | 2-4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada